CLINICAL TRIAL: NCT01188538
Title: Anti P. Acnes Activity of Epiduo® Gel Compared to Benzoyl Peroxide (BPO) 2.5% Gel in the Treatment of Subjects With Acne Vulgaris
Brief Title: Anti Propionibacterium(P.) Acnes Activity of Epiduo® Gel Compared to Benzoyl Peroxide (BPO) 2.5% Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.03.SPR.29084
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2011-07-07 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2011-07

CONDITIONS: Acne Vulgaris
Keywords: P. acnes, Acne vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epiduo gel (Experimental): * Dose or Concentration:Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel.
  * Mode and Frequency of Administration:Topical to the face, once daily application in the evening.
  * Duration of Treatment:12 weeks
  Interventions: Drug: Epiduo gel
- BPO gel (Active Comparator): * Dose or Concentration:Adapalene 0% / Benzoyl Peroxide 2.5% Gel.
  * Mode and Frequency of Administration:Topical to the face, once daily application in the evening.
  * Duration of Treatment:12 weeks
  Interventions: Drug: BPO

INTERVENTIONS:
Drug: Epiduo gel — Once daily application on the face in the evening for 12 weeks
  Other Names: Epiduo
  Arms: Epiduo gel
Drug: BPO — Once daily application on the face in the evening for 12 weeks
  Arms: BPO gel

SUMMARY:
The purpose of this study is to evaluate the antibacterial activity of Epiduo® Gel (Adapalene 0.1% / Benzoyl Peroxide 2.5% Gel) on P. acnes compared to that of Benzoyl Peroxide 2.5% Gel.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with facial acne,
* Subjects with high levels of P. acnes counts on the forehead

Exclusion Criteria:

* Female Subjects who are pregnant, nursing or planning a pregnancy during the study,
* Subjects with acne conglobata, acne fulminans, secondary acne
* Subjects with known or suspected allergy to one of the test product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej LANGNER, Professor, Principal Investigator — Dermatologiczna Klinika Uzdrowiskowa, IWOLANG Sp. z o.o. , Zespół Naukowo-Kliniczny, IWONICZ ZDRÓJ - POLAND
Locations (1):
- Dermatologiczna Klinika Uzdrowiskowa, Iwonicz-Zdrój, Poland

REFERENCES:
- See also: Related Info — http://www.galderma.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 patients have been enrolled in one site in Poland: First subject included: March 3, 2010; last subject out: August 23, 2010
Period: Overall Study
Arm/Group | Epiduo Gel | Benzoyl Peroxide (BPO) Gel
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epiduo Gel | Benzoyl Peroxide (BPO) Gel | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (4.5) | 21.4 (2.9) | 22.1 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 34
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  Poland | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Log10 Cfu/cm²) in Count of Follicular P. Acnes
Description: Quantitative bacterial examinations were performed on the subjects' face during the study. These samplings were performed using a method to quantify the follicular microbiological flora of the skin (at Baseline and Week 12 visits).This method consists of a technique allowing the extraction of the outermost layer of epidermis from hair follicle on the cheek and to culture the samplings in order to have the number of P. acnes.
  Outcome measure = Change from baseline (Log10 cfu/cm²) in count of Follicular P. acnes at end of the study.
Time Frame: Week 12
Population: Intent To Treat (ITT)/Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Log10 cfu/cm²
Arm/Group | Epiduo Gel | Benzoyl Peroxide (BPO) Gel
Number analyzed (Participants) | 20 | 20
Log10 cfu/cm² | -1.94 (1.69) | -1.56 (1.25)

2. Secondary Outcome: Percent Change (%) in Inflammatory Lesion Counts
Description: Inflammatory lesions were counted and recorded by the Evaluator (Investigator or designee) at Baseline and at Week 12. Based on these counts at Baseline and Week 12, Percent change (%) from Baseline in inflammatory lesion counts at Week 12 was calculated.
Time Frame: Week 12
Population: ITT (LOCF)
Measure: Median (Full Range); unit: Percent change (%)
Groups:
- Epiduo® Gel: Epiduo® Gel Topical to the face, once daily application in the evening
- BPO Gel: BPO Gel Topical to the face, once daily application in the evening
Arm/Group | Epiduo® Gel | BPO Gel
Number analyzed (Participants) | 20 | 20
Percent change (%) | -62.8 [-93.3 to 11.1] | -68.1 [-100 to 11.1]

ADVERSE EVENTS:
Time Frame: During the study (from baseline to Week 12)
Description: Questioning at each follow up visit
Arm/Group | Epiduo Gel | Benzoyl Peroxide (BPO) Gel
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Epiduo Gel (N=20) | Benzoyl Peroxide (BPO) Gel (N=20)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other